CLINICAL TRIAL: NCT03898401
Title: Effect of PRP Injection in Releiving of Symptoms of Senile Vaginitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Principal Investigator, rasha medhat abdul-hady, Clinical professor, Ain Shams University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2455
Record Dates: First submitted 2019-03-19; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Senile Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (30):
- 1 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 2 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 3 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 4 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 5 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 6 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 7 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 8 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 9 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 10 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 11 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 12 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 13 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 14 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 15 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 16 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 17 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 18 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 19 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 20 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 21 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 22 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 23 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 24 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 25 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 26 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 27PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 28 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 29 PRP (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma
- 30 PRp (Experimental): Inclusion criteria:
  I. Postmenopausal for at least 3 years. II. Vaginal health index <15. III. Any parity.
  Exclusion criteria:
  I. Women with vaginal infection. II. Women taking estrogen therapy for senile vaginitis. III. Any patient with medical disorder especially diabetes mellitus. IV. Previous vaginal surgery as fistula repair or classical repair. V. Vaginal prolapse VI. Any patient taking chemo or radiotherapy.
  Interventions: Combination Product: Platelet rich plasma

INTERVENTIONS:
Combination Product: Platelet rich plasma — After isolation of the PRP, calcium chloride (0.5ml) was added to the 5 ml of PRP isolate to activate the thrombin cascade, thereby causing degranulation of platelets, releasing growth factors and cytokines, and starting the transformation of the PRP to platelet rich fibrin matrix (PRFM) Before the PRFM became too gelatinous for passing through a needle (less than 10 minutes), two injections will be given through a 27-gauge needle in the posterior vaginal wall and perform clinical evaluations at 0, 1, 3, and 6 months.

SUMMARY:
30 postmenopausal females with senile vaginitis will be enrolled with score of <15 on the Gloria Bachman Vaginal Health Index (VHI) intramucosal injections of PRP will be adminstered and perform clinical evaluations at 0, 1, 3, and 6 months.

DETAILED DESCRIPTION:
30 postmenopausal females with senile vaginitis will be enrolled with score of <15 on the Gloria Bachman Vaginal Health Index (VHI) intramucosal injections of PRP will be adminstered and perform clinical evaluations at 0, 1, 3, and 6 months.

The patients will be seen in Ain shams university gynecological clinic and will not be paid either to receive the procedure or to complete the survey. All patients were fully informed of the innovative therapeutic and experimental nature of the localized PRP injection and consented to the procedure.

The materials and equipment included the following:

1. 5 cc syringes.
2. 27 gauge needles.
3. Centrifuge with proprietary collection system.
4. Calcium chloride 10% (for activation of PRP).
5. and a topical anesthetic cream compounded with a base that prevents irritation and promotes absorption through the vaginal mucosa. Active ingredients will be as follows: bupivicaine, lidocaine, and tetracaine with percent concentrations of 20/8/8 respectively.

First, a topical anesthetic cream will be applied to the posterior vaginal wall. Delaying the PRP injection for 20 minutes after anesthetic application achieved complete or near complete analgesia for the procedure. Peripheral blood will be drawn from the arm and centrifuged to yield 5 cc of PRP. The Regen® system concentrates 5ml of PRP from 10 ml of whole blood using a gel separator.

Study Interventions:

After isolation of the PRP, calcium chloride (0.5ml) was added to the 5 ml of PRP isolate to activate the thrombin cascade, thereby causing degranulation of platelets, releasing growth factors and cytokines, and starting the transformation of the PRP to platelet rich fibrin matrix (PRFM) Before the PRFM became too gelatinous for passing through a needle (less than 10 minutes), two injections will be given through a 27-gauge needle in the posterior vaginal wall and perform clinical evaluations at 0, 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal for at least 3 years.
* Vaginal health index <15.
* Any parity.

Exclusion Criteria:

* Women with vaginal infection.
* Women taking estrogen therapy for senile vaginitis.
* Any patient with medical disorder especially diabetes mellitus.
* Previous vaginal surgery as fistula repair or classical repair.
* Vaginal prolapse
* Any patient taking chemo or radiotherapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of vaginal mucosa using vaginal health index score | 6 months
  Elasticity,fluid volume,integrity,pH,moisture

SECONDARY OUTCOMES:
Female Sexual Distress (FSD) scale | 6 months
  How often did you feel distreesed about your sexual life ?

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Medhat, Professor, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain shams University, Cairo, Elabbasia
  - Ain shams university hospital, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamid ASA, AbdAllah AM, Fathi HM, Eldin AMB, Abd El Hadi RMM. Value of injection of plasma-rich platelets in the vaginal mucosa in cases with vulvovaginal atrophy: a prospective double-blinded randomized controlled study. BMC Womens Health. 2025 Nov 25;25(1):576. doi: 10.1186/s12905-025-04076-5. PMID 41291715